CLINICAL TRIAL: NCT01066208
Title: ACR/EULAR Endorsed Study to Develop New Diagnostic and Classification Criteria for Primary Systemic Vasculitis
Brief Title: American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Diagnostic and Classification Criteria for Primary Systemic Vasculitis
Acronym: DCVAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: American College of Rheumatology (Other); The European League Against Rheumatism (EULAR) (Unknown); The Vasculitis foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACREULAR001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Wegener's Granulomatosis; Microscopic Polyangiitis; Churg Strauss Syndrome; Polyarteritis Nodosa; Giant Cell Arteritis; Takayasu Arteritis
Keywords: Classification criteria; Diagnostic criteria
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa; Giant Cell Arteritis; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients may be given the option of having blood, urine or other tissue obtained as part of their routine care retained for use in future ethically approved studies. They may also be asked to provide additional blood to be stored for this purpose. This component is an optional extra, and does not form part of the main study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (14):
- WG classification: Patients with Wegener's granulomatosis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- MPA classification: Patients with microscopic polyangiitis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- CSS classification: Patients with Churg Strauss syndrome. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- PAN classification: Patients with polyarteritis nodosa. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- Control Classification: For each of the diseases being evaluated (WG, MPA, CSS, PAN, GCA, TAK), patients with the other 5 diseases will be the control group. Within these groups, 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- WG diagnostic: Patients with a new presentation of Wegener's granulomatosis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- MPA diagnostic: Patients with a new presentation of microscopic polyangiitis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- CSS diagnostic: Patients with a new presentation of Churg Strauss syndrome. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- PAN diagnostic: Patients with a new presentation of polyarteritis nodosa. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- Control diagnostic: Patients without vasculitis, but presenting with similar features to the 6 different types of vasculitis being studied. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- GCA classification: Patients with giant cell arteritis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- TAK classification: Patients with Takayasu arteritis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Classification criteria.
- GCA diagnostic: Patients with a new diagnosis of giant cell arteritis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.
- TAK diagnostic: Patients with a new diagnosis of Takayasu arteritis. 1st half of these patients will be assigned to the development cohort and the second half to the validation cohort. Diagnostic criteria.

SUMMARY:
Vasculitis is group of diseases where inflammation of blood vessels is the common feature. Patients typically present with fever, fatigue, weakness and muscle and joint aches. These symptoms are very common among many different diseases, not just vasculitis. A clustering of other symptoms, physical examination findings, blood tests, radiology and biopsy help make the diagnosis. There are currently no criteria to help doctors make a diagnosis of vasculitis when a patient presents with these non specific symptoms and they are reliant on previous experience and disease definitions. One of the aims of this project is to develop diagnostic criteria for the primary systemic vasculitides (granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis, Churg Strauss syndrome, polyarteritis nodosa, giant cell arteritis, Takayasu arteritis). We, the investigators, will do this by studying a large group of patients with vasculitis and comparing them to a large group of patients that present in a similar way, but do not have vasculitis. By comparing the 2 groups we will create a list of items to differentiate between vasculitis and 'vasculitis mimics'.

We also aim to update the current classification criteria. Classification criteria are used to group patients into different types of vasculitis, once a diagnosis of vasculitis has been made, and are useful for studying patients in clinical trials with similar or identical diseases. The current classification criteria (American college of Rheumatology 1990 criteria) were developed 20 years ago, before the availability of some important diagnostic tests (e.g. antineutrophil cytoplasmic antibodies [ANCA]), and are now not consistent with some of the current disease definitions. Therefore to progress future research in vasculitis, it is important that the classification criteria are updated. We will recruit 260 patients with each of the 6 types of vasculitis and compare them with 1300 controls (patients with the 5 other types of vasculitis), in order to determine the optimal combination of symptoms, signs and investigations that classify each person into the appropriate group.

DETAILED DESCRIPTION:
The systemic vasculitides are a group of uncommon but important diseases whose prognosis has improved dramatically with the use of immunosuppressive therapy. However, long-term morbidity from recurrent disease flares, low-grade grumbling disease and/or accumulating damage from previous disease activity or drug therapy now characterise the long-term outlook for patients with vasculitis. There remains major controversy, and incompatibility between the ANCA-associated vasculitides: granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis, and Churg Strauss Syndrome, as well as polyarteritis nodosa in the current classification criteria and disease definitions. Importantly, there are no diagnostic criteria for any of the primary systemic vasculitides.

We propose to improve existing classification criteria for the primary systemic vasculitides. As a starting point will include the following diseases: granulomatosis with polyangiitis (Wegener's) (GPA), microscopic polyangiitis (MPA), Churg Strauss syndrome (CSS), polyarteritis nodosa (PAN), giant cell arteritis (GCA) and Takayasu arteritis (TAK).

We propose to develop and validate classification and diagnostic criteria for primary systemic vasculitis using the guidelines suggested by the Classification and Response Criteria Subcommittee of the American College of Rheumatology Committee on Quality Measures. For all patients, a detailed medical history, physical examination, laboratory tests (including ANCA), radiology (including angiography), biopsy results, treatment, Birmingham Vasculitis Activity Score (BVAS)version 3, Vasculitis Damage Index (VDI), will be collected. The exact list of items to be recorded will be determined by the expert panel at the start of the study.

Classification criteria

We will study a minimum of 100 patients (new and existing patients) prospectively within each currently defined disease category (GPA, CSS, MPA, PAN, GCA, TAK) for the development of the classification criteria. We anticipate the need to recruit 130 patients to account for misdiagnosis and dropout to achieve the target of 100 with the confirmed reference diagnosis. This will include patients that have vasculitis which are assumed to be related to ANCA but do not fulfil the current definitions of any of the diseases, and patients with large vessel vasculitis which do not fulfil current definition for GCA or TAK. Therefore new categories of disease may be created as part of this process and some of the current disease categories may be changed to include or exclude certain patients.

The other diseases will be the controls. The same minimum number of patients will be used to validate the criteria. The 1st 100 patients with a formal reference diagnosis that are recruited for each disease will be used for development of the classification criteria; the next 100 consecutive patients recruited with a confirmed reference diagnosis for each disease will be used to validate the criteria. Again we anticipate the need to recruit 130 patients to account for misdiagnosis and dropout to achieve the 100 target. The majority of cases included will be the same as that used for the development of the diagnostic criteria.

In the absence of an established gold standard, we propose to develop a reference standard. Clinical vignettes using clustering of clinical features and investigations will be constructed from actual cases by the steering group. An expert panel will then be asked to classify each vignette. Hypothetical changes will then be made to components of each clinical vignette and the expert panel will be asked to re classify the case. This process will be repeated multiple times in an attempt to determine what key clinical feature influence the expert panel to change the diagnosis. Using this data driven process, a construct of important clinical features for each disease will be determined by the expert panel. Using this new construct, patients will be classified by the expert panel. This will form the reference standard against which the new criteria will be tested.

Diagnostic Criteria

We propose to develop and validate diagnostic criteria for primary systemic vasculitis. Based on current disease categories we will include GPA, MPA, CSS, PAN, GCA and TAK (but this may change depending on whether new categories are created or existing categories merged as part of the classification criteria component). For the development of diagnostic criteria, we will study a minimum of 100 patients (will require approx 130 patients to allow for dropout and misdiagnosis) for each disease category. Assuming 6 disease categories, the majority of these 780 patients will have already been identified from the classification criteria component of the study and will be re used for the development and validation of diagnostic criteria. However, for the diagnostic criteria to be clinically relevant we will only include patients that are seen at the time of 1st presentation, therefore not all the 780 patients recruited for the classification criteria section of the study will be suitable, and we will need to recruit additional new patients for each of the types of vasculitis being studied.

We will use a minimum of 400 context specific controls (patients that don't have vasculitis) for AAV and PAN that will cover the spectrum of different disease presentations and severity. In addition, we will recruit a minimum of 100 context specific controls for GCA and a similar number for TAK. Different control populations are needed for AAV, GCA and TAK as they have significantly different clinical presentations. In a similar manner to cases, we will recruit 30% more patients than the minimum required to account for misdiagnosis and drop out. The same minimum number of cases and controls will be needed to validate the criteria. The first half of the patients recruited would be used to develop the criteria, and the 2nd half to validate the criteria. We will allow inclusion of patients from previously studied prospective cohorts that meet all the appropriate inclusion / exclusion criteria and have had all the appropriate clinical information and mandatory investigation (to be defined later) recorded at time of their first presentation. This is to facilitate the recruitment of sufficient patients with PAN, CSS and TAK which are rare conditions.

Statistical analysis

We will follow the ACR recommended statistical methods for creating the classification criteria. Patients will have been classified into the different types of vasculitis according to the proposed EULAR/ACR schema by the expert panel or as a vasculitis mimic. The outcomes of interest are binary variables indicating whether or not a patient has been classified as having a particular type of vasculitis, such as GPA, MPA, etc. For each outcome, multivariable logistic regression modeling will be used to identify predictors of outcome based on the list of potential predictor variables described earlier. We will also explore the use of Classification And Regression Tree (CART) analysis. This is a tree-building technique ideally suited to the generation of clinical decision rules. Unlike conventional regression methods, patients are partitioned ("split") into different groups based on an exhaustive search of all possible predictor variables. The advantage of CART analysis over conventional methods is that it is non-parametric, so no assumptions are made about the underlying distribution of predictor variables. CART can handle many hundreds of possible predictor variables and can uncover complex interactions between predictors which may be difficult or impossible to uncover using traditional multivariate techniques that can suffer from model over fitting. In addition, clinicians generally do not think in terms of probability but rather in terms of categories, such as low versus high risk. Clinical decision rules generated using CART analysis are more likely to make clinical sense, and hence more likely to be followed in clinical practice.

Once the best items are identified, the expert panel will decide on the best short list of items to be included in each criteria and also choose the most appropriate decision tree. This will provide the best content validity.

The statistical methods to be used for diagnostic criteria will be very similar to that used for the classification criteria. The binary outcome for analysis is whether the person is a case or control (without vasculitis). We repeat the analyses for each of each type of vasculitis e.g. WG versus controls, then CSS versus controls etc

ELIGIBILITY:
Inclusion Criteria for Classification criteria:

1. Adult patients aged >18 years. There is no upper age limit.
2. Ability to give informed consent. If the patient is unable to give informed consent as a result of death or physical incapacity, then informed assent from next of kin.
3. Presumed diagnosis of a primary systemic vasculitis.

Exclusion criteria for classification criteria:

1. Patients < 18 years of age.
2. Inability to provide informed consent.
3. Hepatitis B or C
4. Co-morbidities that explain the clinical symptoms and signs on which the diagnosis of vasculitis is made. E.g. infection, tumour, other inflammatory condition, etc.

Inclusion criteria for diagnostic criteria:

1. Adult patients aged >18 years. There is no upper age limit.
2. Ability to give informed consent. If the patient is unable to give informed consent as a result of death or physical incapacity, then informed assent from next of kin.
3. Suspected diagnosis of a primary systemic vasculitis

Inclusion criteria for controls group for diagnostic criteria:

1. Adult patients aged >18 years. There is no upper age limit.
2. Ability to give informed consent. If the patient is unable to give informed consent as a result of death or physical incapacity, then informed assent from next of kin.
3. Patients presenting to secondary care with one of the following clinical presentations: I.Multi-system disease. Presentation of disease with at least 2 organs involved. II.Pulmonary-renal syndrome. Defined as haemoptysis / pulmonary haemorrhage with acute renal impairment. III.Acute renal failure IV.Acute respiratory distress. V.Chronic upper airways symptoms and signs. VI.Inflammatory polyarthritis. VII.Fever of unknown origin. VIII.Acute or chronic abdominal pain IX.Hypertension. X.Referred to secondary care with suspicion of vasculitis but confirmed not to have vasculitis. XII.New onset headache. XIII.Jaw or tongue pain. XIV.Sudden visual loss. XV.Limb claudication. XVI.Aortic aneurysm >5cm.

Exclusion Criteria for diagnostic criteria:

1. Patients under the age of 18
2. Patient or next of kin unable or unwilling to provide informed consent or assent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary systemic vasculitis or a mimic of these diseases seen in participating secondary or tertiary care centres in Europe, USA, Mexico, Japan, Asia, Australasia.
Sampling Method: Non-Probability Sample
Enrollment: 3588 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Develop new diagnostic and classification criteria for ANCA associated vasculitis and polyarteritis nodosa | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Raashid A Luqmani, DM, FRCP(E), Principal Investigator — University of Oxford, United Kingdom; Peter Merkel, MD, MPH, Principal Investigator — University of Pennsylvania; Richard Watts, DM, FRCP, Principal Investigator — University of East Anglia
Locations (120):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, LA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Maryland, Baltimore, Maryland
  - Vasculitis Center, Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Internal Medicine, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Centre, Lebanon, NH, Lebanon, New Hampshire
  - New York University Langone Medical Centre, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University Medical Center, Salt Lake City, Utah
- Argentina (2):
  - Hospital Interzonal San Juan Bautista, Catamarca, Catamarca Province
  - Ramos Mejia Hospital, University of Buenos Aires, Buenos Aires
- Australia (2):
  - ANU Medical Centre, Canberra, Australian Capital Territory
  - Royal Brisbane and Women's Hospital, Herston, Queensland
- Medical University Innsbruck, Innsbruck, Austria
- University Hospitals Leuven, Leuven, Belgium
- Canada (8):
  - University of Manitoba, Winnipeg, Manitoba
  - St Joseph's Healthcare, Hamilton, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - Sherbrooke University Hospital Centre, Sherbrooke, Quebec
  - University of Calgary, Calgary
  - St Joseph's Healthcare London, Ontario, Ontario
- Peking Union Medical College Hospital, Beijing, Beijing, China
- Czechia (2):
  - General University Hospital, Prague, Prague
  - General University Hospital, Prague
- Rigshospitalet, Copenhagen, Denmark
- Egypt (2):
  - Assiut University, Assiut University Hospitals, Asyut
  - Cairo University, Kasr El Ainy Hospital, Cairo
- Helsinki University Central Hospital, Helsinki, Finland
- Cochin Hospital, Université Paris-descartes, Paris, France
- Germany (5):
  - Universitätsklinikum Münster, Münster, Münster
  - Universitätsklinikum Jena, Jena
  - University of Schleswig-Holstein, Lübeck
  - Kreiskliniken Esslingen, Plochingen
  - University Hospital Tübingen, Tübingen
- University of Debrecen Medical and Health Science Center, Debrecen, Hungary
- India (5):
  - Chatrapathi Shahuji Maharaj Medical Center, Lucknow (IProcess), Lucknow, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh
  - Nizam's Institute of Medical Sciences, Hyderabad, Hyderabad
  - Medanta, Delhi, New Delhi
  - Christian Medical College & Hospital, Vellore, Vellore
- Ireland (2):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin, Dublin
- Italy (3):
  - University of Parma, Parma
  - Santa Maria Nuova Hospital, Reggio Emilia, Reggio Emilia
  - Arcispedale Santa Maria Nuova, Reggio Emilia
- Japan (14):
  - Kameda Medical Centre, Kamogawa, Kamogawa, Chiba
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Miyazaki University Hospital, Miyazaki, Miyazaki
  - Saitama Medical University, Kawagoe, Saitama
  - Kyorin University Hospital, Mitaka, Tokyo
  - Chiba University, Chiba
  - Kagawa University Hospital, Kagawa
  - St. Marianna University Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - Okayama University Hospital, Okayama
  - Kitano Hospital, Osaka
  - Juntendo University Koshigaya Hospital, Saitama
  - Jichi Medical University Hospital, Tochigi-ken
  - University Tokyo Hospital, Tokyo
- Mexico (2):
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
- New Zealand (4):
  - University of Otago, Christchurch, Christchurch, Canterbury
  - Auckland District Health Board, Auckland
  - Waitemata District Health Board, North Shore Hospital, Auckland
  - Waikato District Health Board, Hamilton
- Norway (2):
  - Hospital of Southern Norway, Kristiansand
  - The University Hospital of Northern Norway, Tromsø, Tromsø
- University of Jagiellonian, Krakow, Poland
- Portugal (3):
  - Hospital Garcia de Orta, Almada, Almada
  - Santa Maria Hospital, Lisbon, Lisbon
  - Hospital Santo Antonio, Porto, Porto
- First Moscow State Medical University, Moscow, Russia
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Seoul National University Hospital, Seoul, South Korea
- Clinic Barcelona Hospital Universitari, Barcelona, Catalonia, Spain
- University of Colombo, Colombo, Sri Lanka
- Sweden (5):
  - Lund University, Lund, Lund
  - Karolinska Institute, Stockholm, Stockholm
  - Linköping University, Stockholm
  - Umeå University, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (2):
  - University Hospital Basel, Basel
  - Immunologie-Zentrum Zurich, Zurich
- Turkey (Türkiye) (6):
  - Hacettepe University, Ankara
  - Istanbul University, Cerrahpasa Medical School, Istanbul
  - Marmara University Medical School, Istanbul
  - Fatih University Medical Faculty, Istanbul
  - Haydarpasa Education and Research Hospital, Istanbul
  - Istanbul University, Istanbul Medical School, Istanbul
- United Kingdom (22):
  - North Cumbria University Hospitals, The Cumberland Infirmary, Carlisle, Cumbria
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - Queen's Hospital, Romford, Essex
  - Southend University Hospital NHS Trust, Westcliff-on-Sea, Essex
  - NHS Fife, Whyteman's Brae Hospital, Windygates, Kirkcaldy, Fife
  - Norfolk and Norwich University Hospital, Norwich, Norwich
  - Nuffield Orthopaedic Centre, Oxford, Oxford
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - NHS Greater Glasgow & Clyde, Gartnavel Hospital, Glasgow, Scotland
  - Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton, Surrey
  - University of Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Dudley Group of Hospitals, NHS FT, Dudley
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University of Manchester, Manchester Royal Infirmary, Manchester
  - Nottingham University Hospitals NHS Trust (QMC), Nottingham
  - Oxford University Hospitals NHS Trust (The Churchill Hospital), Oxford
  - Royal Berkshire NHS Trust, Reading
  - Heatherwood & Wexham Park Hospitals NHS Foundation Trust, Slough
  - Southampton University Hospitals NHS Trust, Southampton
  - York Hospital NHS Foundation Trust, York

REFERENCES:
- [Background] Singh JA, Solomon DH, Dougados M, Felson D, Hawker G, Katz P, Paulus H, Wallace C; Classification and Response Criteria Subcommittee of the Committee on Quality Measures, American College of Rheumatology. Development of classification and response criteria for rheumatic diseases. Arthritis Rheum. 2006 Jun 15;55(3):348-52. doi: 10.1002/art.22003. PMID 16739201
- [Background] Rao JK, Allen NB, Pincus T. Limitations of the 1990 American College of Rheumatology classification criteria in the diagnosis of vasculitis. Ann Intern Med. 1998 Sep 1;129(5):345-52. doi: 10.7326/0003-4819-129-5-199809010-00001. PMID 9735061
- [Background] Hunder GG, Arend WP, Bloch DA, Calabrese LH, Fauci AS, Fries JF, Leavitt RY, Lie JT, Lightfoot RW Jr, Masi AT, et al. The American College of Rheumatology 1990 criteria for the classification of vasculitis. Introduction. Arthritis Rheum. 1990 Aug;33(8):1065-7. doi: 10.1002/art.1780330802. No abstract available. PMID 2390119
- [Background] Fries JF, Hunder GG, Bloch DA, Michel BA, Arend WP, Calabrese LH, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of vasculitis. Summary. Arthritis Rheum. 1990 Aug;33(8):1135-6. doi: 10.1002/art.1780330812. No abstract available. PMID 2202312
- [Background] Jennette JC, Falk RJ, Andrassy K, Bacon PA, Churg J, Gross WL, Hagen EC, Hoffman GS, Hunder GG, Kallenberg CG, et al. Nomenclature of systemic vasculitides. Proposal of an international consensus conference. Arthritis Rheum. 1994 Feb;37(2):187-92. doi: 10.1002/art.1780370206. PMID 8129773
- [Background] Sorensen SF, Slot O, Tvede N, Petersen J. A prospective study of vasculitis patients collected in a five year period: evaluation of the Chapel Hill nomenclature. Ann Rheum Dis. 2000 Jun;59(6):478-82. doi: 10.1136/ard.59.6.478. PMID 10834866
- [Background] Felson DT, Anderson JJ. Methodological and statistical approaches to criteria development in rheumatic diseases. Baillieres Clin Rheumatol. 1995 May;9(2):253-66. doi: 10.1016/s0950-3579(05)80189-x. PMID 7656339
- [Derived] Yates M, MacGregor AJ, Robson J, Craven A, Merkel PA, Luqmani RA, Watts RA. The association of vascular risk factors with visual loss in giant cell arteritis. Rheumatology (Oxford). 2017 Apr 1;56(4):524-528. doi: 10.1093/rheumatology/kew397. PMID 27940595
- See also: Website for European Vasculitis Study Group (EUVAS) — http://www.vasculitis.org